CLINICAL TRIAL: NCT03180905
Title: ImPACT Normative Extension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImPACT Applications, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: QPR-17-03
Record Dates: First submitted 2017-05-23; First posted 2017-06-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Validity (Experimental): ImPACT Online a computerized test will be administered to subjects. They will also receive a battery of paper and pencil neuropsychological tests.
  Interventions: Device: ImPACT Online/Paper Pencil Tests
- Test/Re-Test (Active Comparator): ImPACT Online will be administered at 2 time points
  Interventions: Device: ImPACT Online

INTERVENTIONS:
Device: ImPACT Online/Paper Pencil Tests — Compare ImPACT Online versus Paper and Pencil Neurocognitive Tests
  Arms: Validity
Device: ImPACT Online — ImPACT Online will be administered at 2 time points.
  Arms: Test/Re-Test

SUMMARY:
The researchers want to find out more about a standalone software application, ImPACT Online and how it relates to other commonly used tests of memory, attention and reaction time. ImPACT Online is a computer-based neurocognitive test for concussion management. The test was designed to help measure the effects of concussion on cognitive processes (for example, memory, attention, brain speed) and visual functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 60-80
2. Primary English speaking or fluent in English.
3. Currently does not reside in a skilled nursing facility.
4. Currently not suffering from a concussion or being treated for a concussion, unless enrolled in the subgroup Discriminative Validity.
5. No known physical, neurological, behavioral or psychological impairment that would affect their ability to perform the test.
6. Hearing or vision impairments that have not been corrected within normal limits.
7. A score of 24 or greater on the MMSE (Mini-Mental State Examination).

Exclusion Criteria:

1. English is not their primary language nor are they proficient in the English language.
2. Currently resides in a skilled nursing facility.
3. Currently suffering from a concussion or being treated for a concussion, unless enrolled in the subgroup Discriminative Validity.
4. Known physical, neurological, behavioral, or psychological impairment that would affect their ability to take or complete the test.
5. Hearing or vision impairments that would affect their ability to perform the test.
6. Score of 23 or below on the MMSE(Mini-Mental State Examination).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity | 12 Months
  ImPACT Online compared to Brief Visuospatial Memory Test
Validity | 12 Months
  ImPACT Online compared to Symbol Digit Modalities Test
Validity | 12 Months
  ImPACT Online compared to Color Trails
Validity | 12 Months
  ImPACT Online compared to Hopkins Verbal Learning Test.

SECONDARY OUTCOMES:
Reliability | Baseline Test will be administered at enrollment and re- test will be administered within 30 days of baseline test.
  Reliability will be established through a test/re-test. Online ImPACT will be administered at 2 time points to establish results should be stable over time.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Comprehensive Med Psych Systems, Inc., Sarasota, Florida
  - University of Albany, Albany, New York
  - ImPACT Applications Inc., Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No